CLINICAL TRIAL: NCT02973360
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Finding Study and Open-Label Extension of SC411 in Children With Sickle Cell Disease
Brief Title: Dose-Finding Study of SC411 in Children With Sickle Cell Disease
Acronym: SCOT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Micelle BioPharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMEG-411-02
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Docosahexaenoic Acids; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 (Experimental): Target dose 20 mg/kg Docosahexaenoic acid
  Interventions: Drug: Docosahexaenoic Acid
- Dose Level 2 (Experimental): Target dose 36 mg/kg Docosahexaenoic acid
  Interventions: Drug: Docosahexaenoic Acid
- Dose Level 3 (Experimental): Target dose 60 mg/kg Docosahexaenoic acid
  Interventions: Drug: Docosahexaenoic Acid
- Placebo (Placebo Comparator): Soybean oil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Docosahexaenoic Acid — Oral Capsule
  Other Names: SC411
  Arms: Dose Level 1; Dose Level 2; Dose Level 3
Drug: Placebo — Oral Capsule
  Other Names: Soybean oil
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group, dose-finding study of SC411 in children with sickle cell disease (SCD). The primary objective of the study is to evaluate the safety and tolerability of three different doses of SC411 compared to a placebo. All patients will undergo eight weeks of oral study treatment and a four-week safety follow-up period. Patients will be randomized to one of three dose levels of SC411 or placebo.

DETAILED DESCRIPTION:
This Phase 2 study is to be conducted in two parts. Part A is a randomized, double-blind, placebo-controlled, parallel-group, dose-finding study of SC411 in children with SCD. This part of the study will consist of a screening period of up to 2 weeks, followed by an eight-week treatment period. Part B is an optional 49-month open-label extension for patients who have completed Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than or equal to 5 years and less than or equal to 17 years at screening;
2. Has been diagnosed with SCD that includes the phenotypes HbSS, hemoglobin SC, and HbS/beta-thalassemia. Hemoglobin phenotyping must be previously documented by either hemoglobin high-performance liquid chromatography [HPLC] or electrophoresis at time of Screening. If a patient does not have documented hemoglobin phenotyping at the time of Screening, or has received a blood transfusion within the two months prior to the Screening Visit, hemoglobin phenotyping should be documented by hemoglobin HPLC;
3. Has had at least two and no more than ten documented episodes of clinical sickle cell crises within 12 months prior to the Screening Visit. A sickle cell crisis is defined as an episode of vaso-occlusive event:

   * Painful crisis defined as new onset of pain that lasts two or more hours for which there is no explanation other than vaso-occlusion, and which requires therapy with oral or parenteral opioids, non-steroidal anti-inflammatory drugs, or other analgesics prescribed by a healthcare provider in a medical setting such as a hospital, clinic, or emergency room visit, or documented telephone management (Ballas, 2010; Heeney, 2016; Jacob, 2005); and
   * Acute chest syndrome defined as acute illness characterized by a new segmental pulmonary infiltrate on a chest x-ray, and fever (greater than or equal to 38.5°C) or respiratory symptoms such as hypoxia, chest pain, tachypnea, wheezing, or cough (Ballas, 2010);
4. Is either not on hydroxyurea at the Screening Visit and does not plan on receiving it during the course of the first 12 weeks of the study (Part A), or has received hydroxyurea for a minimum of 6 months and, except for safety reasons, will remain on the same weight-based dose of hydroxyurea from screening throughout the duration of Part A of the study;
5. Parent or guardian is able to give written informed consent, and the potential pediatric patient is able to provide assent in a manner approved by the Institutional Review Board (IRB) and comply with the requirements of the study other than for safety reasons; and
6. If sexually active, agrees to use a reliable method of birth control (eg, barrier, birth control pills, abstinence) during the study and for one month following the last dose of study drug.

Exclusion Criteria:

1. Has a significant medical condition that required hospitalization (other than sickle cell crisis) within two months of the Screening Visit;
2. Has a known allergy or hypersensitivity to fish or shellfish;
3. Has a known allergy or hypersensitivity to soy;
4. Is planning to initiate, terminate, or alter the dosing of hydroxyurea during the first 12 weeks of the study, other than for safety reasons;
5. Has chronic daily use (more than 30 consecutive days during the last six months prior to enrollment) of opioid analgesia for any reason;
6. Has a diagnosis of chronic pain or chronic pain syndrome (eg, chronic pain from the repeated vaso-occlusive events, chronic pain from avascular necrosis);
7. Has a history of Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C infection;
8. Has a history of documented episode(s) of priapism within 12 months of the Screening Visit;
9. Has a history of atrial or ventricular arrhythmia;
10. Has an international normalized ratio (INR) >2.0, or is on regular anticoagulation therapy, or has a history of a known bleeding diathesis;
11. Has thrombocytopenia (platelets less than 80,000) or is on chronic acetylsalicylic acid therapy;
12. Has increased risk of stroke: documented abnormal or "high conditional" transcranial Doppler (TCD) mean velocity (TCD V) by STOP criteria (Adams, 1998) within the preceding year or has a history of known cerebrovascular disease:

    * "High conditional" = TCD V greater than or equal to 185 to 199 cm/sec, or TCDi V greater than or equal to 170 to 184 cm/sec, or TCD maximum V greater than or equal to 250 cm/sec; or
    * Abnormal = TCD V greater than or equal to 200 cm/sec, or abnormal high TCDi V greater than or equal to 185 cm/sec, or TCD maximum V greater than or equal to 250 cm/sec;
13. Has received a blood transfusion or exchange transfusion in the three months prior to the Screening Visit;
14. Has renal insufficiency (creatinine greater than 1.5 times upper limit of normal [ULN], or requiring peritoneal dialysis or hemodialysis);
15. Has liver dysfunction (ALT greater than 2.0 times ULN);
16. Has other concomitant chronic medical or psychiatric condition that, in the opinion of the Investigator, would compromise participation in the study or confound the evaluation of the study outcome;
17. Is pregnant or lactating or has the intention of becoming pregnant during the study (if a female of child-bearing potential or partner of a patient participating in the study);
18. Is currently taking, or has been treated with, any form of omega-3 fatty acid or fish oil supplement within 30 days of the Screening Visit or during the course of the study;
19. Has been treated with an experimental anti-sickling medication/treatment within 30 days of the Screening Visit or during the course of the study;
20. Is currently taking or has been treated with any investigational drug for any disease within 30 days of the Screening Visit or during the course of the study;
21. Is currently enrolled in an investigational drug or device study and/or has participated in such a study within 30 days of the Screening Visit or during the course of the study; or
22. There are factors that would, in the judgment of the Investigator, make it difficult for the patient to comply with the requirements of the study (eg, inability to swallow capsules due to past history of stroke, or poor compliance).

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2022-01-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety & tolerability of SC411 & determine change from Baseline in the blood cells omega-3 fatty acids index in subjects, treated with active SC411 doses or placebo in Part A and safety and tolerability in Part B. | Week 0 (baseline) through Month 52 (end of treatment)
  Evaluate the safety and tolerability of three different doses of SC411 and determine the change from Baseline in the blood cells omega-3 fatty acids index in subjects, treated with either one of the three active doses of SC411 or matching placebo in Part A. Safety and tolerability will continue to be evaluated and reported during Part B.

SECONDARY OUTCOMES:
Measurement of the pharmacokinetic (PK) parameter of AUC will be performed for three dose levels of SC411 will be measured. | 2 weeks before baseline (screening) through Week 52
  Measurement of the pharmacokinetic (PK) parameter of AUC will be performed for three dose levels of SC411 will be measured.
  The steady-state pharmacokinetic (PK) profile of the three doses and area under the curve will be reported. The purpose is to assess the steady-state pharmacokinetic (PK) profile of the three dose levels of SC411, following two months of dosing, and at the end of treatment (EOT).
Measurement of the pharmacokinetic (PK) parameter of Tmax will be performed for three dose levels of SC411 will be measured. | 2 weeks before baseline (screening) through Week 52
  Measurement of the pharmacokinetic (PK) parameter of Tmax will be performed for three dose levels of SC411 will be measured.
  The steady-state pharmacokinetic (PK) profile of the three doses and Tmax will be reported. The purpose is to assess the steady-state pharmacokinetic (PK) profile of the three dose levels of SC411, following two months of dosing, and at the end of treatment (EOT).
Measurement of the pharmacokinetic (PK) parameter of Cmax will be performed for three dose levels of SC411 will be measured. | 2 weeks before baseline (screening) through Week 52
  The steady-state pharmacokinetic (PK) profile of the three doses and Cmax will be reported. The purpose is to assess the steady-state pharmacokinetic (PK) profile of the three dose levels of SC411, following two months of dosing, and at the end of treatment (EOT).
The safety & long term tolerability of SC411 will be evaluated in Part A, & a selected dose in Part B. The change from Baseline in blood cells omega-3 fatty acids index in subjects, treated with SC411 or placebo in Part A will be determined. | Week 0 (baseline) through Month 52 (end of treatment)
  Evaluate the safety and long term tolerability of three different doses of SC411 and determine the change from Baseline in the blood cells omega-3 fatty acids index in subjects, treated with either one of the three active doses of SC411 or matching placebo in Part A. Safety and long term tolerability will continue to be evaluated and reported during Part B.

OTHER OUTCOMES:
The number of painful crises had by subjects receiving one of the three oral dose levels of SC411 compared to matching placebo will be evaluated from eDiary-records of patient reported outcomes. | Week 0 (baseline) through Week 8 plus one day (end of treatment on Part A)
  The exploratory objective of this study are to evaluate the effect of the three oral dose levels of SC411 compared to matching placebo from eDiary-records of patient reported outcomes of painful crises. The number of painful crises will be reported by the patient and evaluated based on SC411 compared to matching placebo.
The intensity of painful crises on a scale of 0 to 10, reported by subjects receiving one of the three oral dose levels of SC411 compared to matching placebo will be evaluated from eDiary-records of patient reported outcomes. | Week 0 (baseline) through Week 8 plus one day (end of treatment on Part A)
  The exploratory objective of this study are to evaluate the effect of the three oral dose levels of SC411 compared to matching placebo from eDiary-records of patient reported outcomes of intensity of painful crises on a scale of 0 to 10, reported by the patient. Painful crises will be reported by the patient and evaluated based on level of intensity.
The number of times the subject reports taking an analgesic at home by subjects receiving one of the three oral dose levels of SC411 compared to matching placebo will be evaluated from eDiary-records of patient reported outcomes. | Week 0 (baseline) through Week 8 plus one day (end of treatment on Part A)
  The exploratory objective of this study are to evaluate the effect of the three oral dose levels of SC411 compared to matching placebo from eDiary-records of patient reported outcomes of the number of times the patient reports taking an analgesic at home. The number of times the patient reports taking an analgesic at home will be reported by the patient and evaluated.
The number of school days missed because of pain by subjects receiving one of the three oral dose levels of SC411 compared to matching placebo will be evaluated from eDiary-records of patient reported outcomes. | Week 0 (baseline) through Week 8 plus one day (end of treatment on Part A)
  The exploratory objective of this study are to evaluate the effect of the three oral dose levels of SC411 compared to matching placebo from eDiary-records of patient reported outcomes of the number of times the patient reports taking an analgesic at home. The number of school days missed because of pain will be reported by the patient and evaluated.
The number of blood transfusions on subjects receiving one of the three oral dose levels of SC411 compared to matching placebo will be evaluated. | Week 0 (baseline) through Week 8 plus one day (end of treatment on Part A)
  The exploratory objectives of this study are to evaluate the effect of the three oral dose levels of SC411 compared to matching placebo on the number of blood transfusions. (acute simple blood transfusions and exchange blood transfusions).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Heeney, MD, Principal Investigator — Boston Children's Hospital
Locations (11):
- United States (11):
  - Children's of Alabama - University of Alabama, Birmingham, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Florida Health at Shands, Gainesville, Florida
  - Batchelor Children's Research Institute - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta - Emory University, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - East Carolina University, Greenville, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Hospital - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daak AA, Dampier CD, Fuh B, Kanter J, Alvarez OA, Black LV, McNaull MA, Callaghan MU, George A, Neumayr L, Hilliard LM, Sancilio F, Rabinowicz AL, Heeney MM. Double-blind, randomized, multicenter phase 2 study of SC411 in children with sickle cell disease (SCOT trial). Blood Adv. 2018 Aug 14;2(15):1969-1979. doi: 10.1182/bloodadvances.2018021444. PMID 30097463
- See also: EFFECTS OF SC411 ON BLOOD CELL MEMBRANE OMEGA-3 INDEX AND SELECT SICKLE CELL DISEASE BIOMARKERS IN THE SCOT TRIAL: A PHASE 2 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP, MULTI-CENTER STUDY — https://aspho.planion.com/Web.User/AbstractDet?ACCOUNT=ASPHO&ABSID=14095&CONF=AM18&ssoOverride=OFF&CKEY
- See also: CLINICAL EFFECT OF SC411 ON CHILDREN WITH SICKLE CELL DISEASE IN THE SCOT TRIAL: A PHASE 2 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP, DOSE-FINDING MULTI-CENTER STUDY — https://aspho.planion.com/Web.User/AbstractDet?ACCOUNT=ASPHO&ABSID=14068&CONF=AM18&ssoOverride=OFF&CKEY